CLINICAL TRIAL: NCT05966948
Title: Hypertonic Dextrose Prolotherapy Versus Normal Saline Intra-articular Injection Among Knee Osteoarthritis With Obese Patient
Brief Title: HDP vs NS Intra-articular Injection Among KOA With Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rumah Sakit Umum Daerah Haji Provinsi Jawa Timur, Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSUHajiJaTimProv
Record Dates: First submitted 2023-07-11; First posted 2023-08-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis; Obesity
Keywords: knee osteoarthritis; obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Glucose; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study involves two arms assigned randomly for receiving different treatment. One arm for Hypertonic Dextrose Prolotherapy as intervention group and Normal Saline as control group.
Who Masked: Participant
Masking Description: Participants who met the eligibility of the study who were on outpatient treatment on that day were randomized in order of queue, odd numbers as the intervention group and even numbers as the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Dextrose Prolotherapy (Experimental): This group received a Hypertonic dextrose intra articular is 25%, while extra articular 20% injection on day 1 and day 30 with same dose.
  Interventions: Drug: Dextrose Solution
- Normal Saline (Placebo Comparator): This group received Normal Saline injection on day 1 and day 30.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dextrose Solution — Prolotherapy is a regenerative tissue therapy that is considered efficacious for reducing the symptoms and morbidity of Knee Osteoarthritis (KOA) using hypertonic dextrose as an injectable substance. Treatment will be given two times, on day 1st and 30th day.
  Other Names: Dextrose Injection
  Arms: Hypertonic Dextrose Prolotherapy
Drug: Normal Saline — Normal Saline will be intra-articular injected and given two times, on day 1st and 30th day.
  Other Names: Normal Saline Injection
  Arms: Normal Saline

SUMMARY:
The aim of this randomized controlled trial study was to compare the effect of intra-articular injection of Hypertonic Dextrose Prolotherapy (HDP) with Normal Saline (NS) in the clinical improvement of knee osteoarthritis (KOA) patients with comorbid obesity. The main questions to be answered are:

* How does the effect of HDP versus NS intra-articular injection compare to the numerical rating score (NRS) in obese KOA patients?
* How does the effect of HDP versus NS intra-articular injection compare to scores of The Western Ontario and McMaster Universities Arthritis Index (WOMAC) in obese KOA patients?
* How does the effect of HDP versus NS intra-articular injection compare to the thickness of the femoral cartilage in obese KOA patients?

Participants who meet the inclusion and exclusion criteria will be randomized based on the order of the outpatient department each day, with odd numbers as the HDP intervention group and even numbers as NS. They received ultrasound-guided intra-articular injections on day 1 and day 30.

Researchers will compare HDP versus NS groups to see which group improves NRS, WOMAC, and femoral cartilage thickness.

DETAILED DESCRIPTION:
This is a randomized controlled study, which recruited KOA patients with obese comorbidity who were treated at the Outpatient Department of Physical Medicine and Rehabilitation at Rumah Sakit Daerah Haji Provinsi Jawa Timur, Surabaya, Indonesia from May to August 2023. The participants were divided into two groups, including HDP versus NS injections.

Each study participant's identity including age, gender, weight, height, and BMI was recorded. Then an evaluation of the NRS, WOMAC score, and femoral cartilage thickness was carried out using ultrasound.

This study assessed using the NRS scale for pain reduction on a scale of 0 to 10 (0 means no pain, while 10 means very pain). The WOMAC Score consists of 24 questions with four scales, namely 0: none, 1: mild, 2: moderate, 3: severe, and 4: very severe. Femoral cartilage thickness scan using ultrasound with millimeter units.

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed with knee osteoarthritis (KOA).
* Patient was diagnosed with obesity.

Exclusion Criteria:

* Patient with a history of knee trauma.
* Patient with a history of knee surgery.
* Patient with a history of intra-articular injection before.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Before intervention, day 1, and day 30 after intervention
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. We classified from 0 to 10, where 0 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
WOMAC Score | Before intervention, day 1, and day 30 after intervention
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 sub-scales:
  (1) Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright; (2) Stiffness (2 items): after first waking and later in the day; (3) Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
Femoral Cartilage Thickness | Before intervention, day 1, and day 30 after intervention
  The ultrasound measurement of femoral cartilage thickness is divided into three sites: medial condyle, intercondylar, and lateral condyle on the right and left sides. This measurement is in millimeters units.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Vivera Pane, MD, PhD, Study Chair — Universitas Nahdlatul Ulama Surabaya
Locations (1):
- Rumah Sakit Umum Daerah Haji Provinsi Jawa Timur, Indonesia, Surabaya, East Java, Indonesia

REFERENCES:
- [Background] Cortez VS, Moraes WA, Taba JV, Condi A, Suzuki MO, Nascimento FSD, Pipek LZ, Mattos VC, Torsani MB, Meyer A, Hsing WT, Iuamoto LR. Comparing dextrose prolotherapy with other substances in knee osteoarthritis pain relief: A systematic review. Clinics (Sao Paulo). 2022 May 17;77:100037. doi: 10.1016/j.clinsp.2022.100037. eCollection 2022. PMID 35594623
- [Background] Topol GA, Pestalardo IG, Reeves KD, Elias F, Steinmetz NJ, Cheng AL, Rabago D. Dextrose Prolotherapy for Symptomatic Grade IV Knee Osteoarthritis: A Pilot Study of Early and Longer-Term Analgesia and Pain-Specific Cytokine Concentrations. Clin Pract. 2022 Nov 14;12(6):926-938. doi: 10.3390/clinpract12060097. PMID 36412676
- [Background] Yu T, Yan S, Chi Z, Zhu D, Cheng P, Li H, Qin S, Zhong G, Ouyang X, Chen R, Jiao L. Comparative efficacy and safety of injection therapies for knee osteoarthritis: A protocol for systematic review and Bayesian network meta analysis. Medicine (Baltimore). 2020 Nov 20;99(47):e22943. doi: 10.1097/MD.0000000000022943. PMID 33217798
- [Background] Sit RWS, Wu RWK, Rabago D, Reeves KD, Chan DCC, Yip BHK, Chung VCH, Wong SYS. Efficacy of Intra-Articular Hypertonic Dextrose (Prolotherapy) for Knee Osteoarthritis: A Randomized Controlled Trial. Ann Fam Med. 2020 May;18(3):235-242. doi: 10.1370/afm.2520. PMID 32393559
- [Background] Pane RV, Setiyaningsih R, Widodo G, Al Hajiri AZZ, Salsabil JR. Femoral Cartilage Thickness in Knee Osteoarthritis Patients and Healthy Adults: An Ultrasound Measurement Comparison. ScientificWorldJournal. 2023 Feb 17;2023:3942802. doi: 10.1155/2023/3942802. eCollection 2023. PMID 36845755
- [Background] Akcay S, Gurel Kandemir N, Kaya T, Dogan N, Eren M. Dextrose Prolotherapy Versus Normal Saline Injection for the Treatment of Lateral Epicondylopathy: A Randomized Controlled Trial. J Altern Complement Med. 2020 Dec;26(12):1159-1168. doi: 10.1089/acm.2020.0286. Epub 2020 Sep 28. PMID 32990454
- [Background] Sit RWS, Wu RWK, Reeves KD, Rabago D, Chan DCC, Yip BHK, Chung VCH, Wong SYS. Efficacy of intra-articular hypertonic dextrose prolotherapy versus normal saline for knee osteoarthritis: a protocol for a triple-blinded randomized controlled trial. BMC Complement Altern Med. 2018 May 15;18(1):157. doi: 10.1186/s12906-018-2226-5. PMID 29764447
- [Background] Wee TC, Neo EJR, Tan YL. Dextrose prolotherapy in knee osteoarthritis: A systematic review and meta-analysis. J Clin Orthop Trauma. 2021 May 20;19:108-117. doi: 10.1016/j.jcot.2021.05.015. eCollection 2021 Aug. PMID 34046305
- [Background] Chen YW, Lin YN, Chen HC, Liou TH, Liao CD, Huang SW. Effectiveness, Compliance, and Safety of Dextrose Prolotherapy for Knee Osteoarthritis: A Meta-Analysis and Metaregression of Randomized Controlled Trials. Clin Rehabil. 2022 Jun;36(6):740-752. doi: 10.1177/02692155221086213. Epub 2022 Mar 8. PMID 35257594
- [Background] Arias-Vazquez PI, Tovilla-Zarate CA, Legorreta-Ramirez BG, Burad Fonz W, Magana-Ricardez D, Gonzalez-Castro TB, Juarez-Rojop IE, Lopez-Narvaez ML. Prolotherapy for knee osteoarthritis using hypertonic dextrose vs other interventional treatments: systematic review of clinical trials. Adv Rheumatol. 2019 Aug 19;59(1):39. doi: 10.1186/s42358-019-0083-7. PMID 31426856